CLINICAL TRIAL: NCT03958773
Title: Cardiovalve Transfemoral Mitral Valve System in Patients at High Surgical Risk With Severe Mitral Regurgitation
Brief Title: Cardiovalve Transfemoral System - FIM Study
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Cardiovalve Ltd. (Industry)
Collaborators: Meditrial Europe Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CP 17-01
Record Dates: First submitted 2019-05-19; First posted 2019-05-22 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Mitral Regurgitation
Keywords: Mitral valve; Functional mitral regurgitation; Heart failure
MeSH Terms: conditions — Mitral Valve Insufficiency; Heart Failure

STUDY DESIGN:
Intervention Model Description: Prospective, single-center, single-arm feasibility clinical study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Cardiovalve treatment (Experimental): Patients that implanted with the Cardiovalve device
  Interventions: Device: Cardiovalve transfemoral Mitral valve system

INTERVENTIONS:
Device: Cardiovalve transfemoral Mitral valve system — Cardiovalve System, comprised of: 1) Cardiovalve Implant; 2) Cardiovalve Delivery System (DS); 3) Cardiovalve Accessories.

SUMMARY:
The Cardiovalve system is a replacement valve delivered through a transfemoral access and transseptal approach and is intended for symptomatic patients with Mitral regurgitation for whom surgical options are not feasible.

DETAILED DESCRIPTION:
The Cardiovalve system is a replacement valve delivered through a transfemoral access and transseptal approach and is intended for symptomatic patients with Mitral regurgitation for whom surgical options are not feasible.

The purpose of this study is to evaluate the safety of the CardiovalveSystem with its associated procedure, and observe the device performance in reducing mitral regurgitation Data collected in this clinical study will include 30-day safety and performance of the device and delivery system, and long-term clinical outcomes over a follow-up of 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* NYHA functional II, III or ambulatory IV
* Severe mitral regurgitation (MR grade 3-4+)
* High risk for conventional open mitral valve repair or replacement surgery in the consideration of the site Heart Team (including a cardiac surgeon, a cardiologist and imaging specialist as a minimum)
* Able to undergo Transesophageal Echocardiography (TEE).
* Subject understands the study requirements and the treatment procedures and provides written Informed Consent before any study-specific tests or procedures are performed.
* The subject commits to return for the scheduled post-operative follow-up visits at the hospital.
* Suitable for femoral access procedure and transseptal catheterization
* Native mitral valve geometry and size and LV outflow tract characteristics compatible with the Cardiovalve

Exclusion Criteria:

* Prior stroke or TIA within 3 months
* Acute myocardial infarction within the previous 30 days
* Any prior heart valve surgery or transcatheter mitral intervention
* Any percutaneous cardiovascular intervention, cardiovascular surgery, or carotid surgery within 30 days
* Rheumatic heart disease or endocarditis within the previous 3 months
* Hypertrophic cardiomyopathy, restrictive cardiomyopathy, constrictive pericarditis, or any other structural heart disease causing heart failure other than dilated cardiomyopathy of either ischemic or non-ischemic etiology
* Existence of inferior vena cava filter or atrial septal device (contraindicating femoral access and transseptal catheterization)
* Untreated clinically significant coronary artery disease requiring revascularization
* Tricuspid valve disease requiring surgery or severe tricuspid regurgitation
* Aortic valve disease requiring surgery Anatomical Exclusion Criteria (assessed by pre-procedural imaging)
* Left Ventricular Ejection Fraction ( LVEF) <30%
* LV end diastolic diameter > 70mm
* Significant abnormalities of the mitral valve and sub-valvular apparatus.
* Severe mitral annular or leaflets calcification
* Left atrial or LV thrombus
* Severe right ventricular dysfunction
* Severe tricuspid or aortic valve disease General Exclusion Criteria
* Subject who is currently participating in an investigational study, other than this study
* Hemodynamic instability defined as systolic pressure < 90mmHg or the need for inotropic support or intra-aortic balloon pump or other hemodynamic support device, or any mechanical heart assistance
* Subject has contrast agent hypersensitivity that cannot be adequately pre-medicated, has an allergy to Nitinol alloys (nickel and titanium), or has intolerance to antiplatelet, anticoagulant, or thrombolytic medications
* Bleeding diathesis or hypercoagulable state
* Active peptic ulcer or active gastrointestinal bleeding
* Pulmonary artery systolic pressure >70 mmHg
* Patients with renal insufficiency (creatinine > 2.5 mg/dL)
* Subject with hepatic insufficiency
* Subject has a co-morbid illness that may result in a life expectancy of less than one year
* Active infection that requires antibiotic therapy
* Subject is pregnant, breastfeeding or intend to become pregnant within one year

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-10-12 (Actual); Primary Completion 2026-10-30 (Estimated); Study Completion 2026-10-30 (Estimated)

PRIMARY OUTCOMES:
Freedom from major device or procedure related serious adverse events | 30 days
  Freedom from major device or procedure related serious adverse events:
  F. Stage 2 or 3 acute kidney injury (includes new dialysis) H. Severe hypotension, worsening of heart failure, or respiratory failure requiring intravenous pressors or invasive or mechanical heart failure treatments such as ultrafiltration or hemodynamic assist devices, including intra-aortic balloon pumps or left ventricular or biventricular assist devices, or prolonged intubation for >48 h.
  I. Any valve-related dysfunction, migration, thrombosis, or other complication requiring surgery or repeat intervention

SECONDARY OUTCOMES:
Technical success | Intraoperative
  Technical success; delivery and deployment of the device in the correct position and retrieval of delivery catheter, without significant mitral stenosis, LVOT obstruction or paravalvular MR documented by intraoperative imaging Number of patients for whom the device was successfully implanted (per MVARC definitions) Number of patients with reduction in MR grade from Baseline Number of patients with improvement in NYHA class from baseline Number of patients with increase distance walked in the 6MW test from baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Rimantas Benetis, MD, Principal Investigator — Head of department
Locations (1):
- Hospital of the Lithuanian University of Health Sciences ligoninė Kauno, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No